CLINICAL TRIAL: NCT01105780
Title: Single Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-41443532 in Healthy Male and Female Caucasian and Male Japanese Subjects
Brief Title: JNJ-41443532 Sex, Race, and Age Pharmacokinetic (PK) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CR017083; 41443532EDI1002 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Healthy; Japanese; Pharmacokinetics; JNJ-41443532
MeSH Terms: interventions — JNJ-41443532

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 001 (Experimental): JNJ-41443532 250mg tablet once daily for 1 day
  Interventions: Drug: JNJ-41443532
- 002 (Placebo Comparator): Placebo Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching placebo
  Arms: 002
Drug: JNJ-41443532 — 250mg tablet once daily for 1 day
  Arms: 001

SUMMARY:
The purpose of this study is to assess the safety, tolerability pharmacokinetics (how the drug is absorbed in the body, how it is distributed within the body and how it is removed from the body over time) and pharmacodynamics (the effects of the drug) of JNJ-41443532 in healthy male and female Caucasian and male Japanese participants.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-controlled, parallel group, single dose study in male and female Caucasian and male Japanese participants. The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) study in healthy male and female caucasian and male Japanese participants. For each participant, the study will consist of a screening examination (within 28 days of first dose on Day 1), a single period of open label treatment (all people involved know the identity of the intervention) upon entry in the study and discharge on Day 3), and a final, follow-up examination between 7-10 days after discharge from the study. Safety assessments include monitoring of adverse events, and evaluation of lab results, cardiac parameters, vital signs, and physical exams. Participants receive study medication (JNJ-41443532 or placebo) by mouth on Day 1 after an overnight fast of at least 10 hours; planned dose is 250 mg.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian or Japanese male
* Japanese participant born in Japan of Japanese parents and maternal and paternal grandparents must not have lived outside of Japan for more than 5 years, and lifestyles including diet, must not have changed significantly since relocating from Japan
* Caucasian male or postmenopausal/surgically sterile Caucasian female
* Caucasian participant born of Caucasian parents and maternal and paternal grandparents must continue their usual lifestyle and diet
* Weight = 50 kilograms and Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 (inclusive)
* Healthy on the basis of physical examination, medical history, vital signs, and electrocardiogram (ECG) and clinical laboratory tests performed at screening
* Men must agree to use a double barrier method of birth control (e.g. condom and use of spermicide with diaphragm, hormonal contraceptives or intrauterine devices by female partner) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Competency in speaking and comprehending the language where the study will be conducted

Exclusion Criteria:

* History of, or currently active, significant illness or medical disorders, including (but not limited to) cardiovascular disease (including cardiac arrhythmias, myocardial infarction, stroke, peripheral vascular disease), endocrine or metabolic disease (e.g. hyper/hypo-thyroidism), hematological disease (e.g. von Willebrand's disease or other bleeding disorders), respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmologic disorders (including retinal disorders or cataracts), neoplastic disease, skin disorder, or any other illness that the Investigator considers should exclude the participant
* Participants at risk for QTc prolongation (specific heart rhythm irregularity)
* Within 12 months prior to screening, has had a clinically important, serious infection (e.g. hepatitis, pneumonia, or pyelonephritis), has been hospitalized for an infection or has been treated with intravenous (IV) antibiotics for an infection
* Smoker or tobacco user within the past 3 months
* History of alcohol or drug abuse
* History of clinically significant drug and/or food allergies, including allergies or intolerance (e.g. lactose intolerance)
* Donation of 1 or more units of blood or acute loss of an equivalent amount of blood within 60 days prior to study drug administration
* Received an experimental drug or used an experimental medical device within 60 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05; Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determine the pharmacokinetic properties of a single dose JNJ-41443532 as determined by blood level concentrations. | 6 Weeks

SECONDARY OUTCOMES:
To explore the pharmacodynamic (PD) effects of JNJ-41443532 and to compare differences in the PD profile by age, sex, and race. | 6 Weeks
To explore the relationship between JNJ-41443532 plasma concentrations (blood levels) and pharmacodynamic effects (concentration-effect relationships). | 6 Weeks
Determine the safety and tolerability of JNJ-41443532 as determined by evaluation of adverse events, lab results, cardiac monitoring, vital signs, and physical exams. | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Cypress, California, United States